CLINICAL TRIAL: NCT03104699
Title: A Phase 1/2, Open-Label, Multiple Ascending Dose Trial to Investigate the Safety, Tolerability, Pharmacokinetics, Biological, and Clinical Activity of AGEN2034 in Subjects With Metastatic or Locally Advanced Solid Tumors, With Expansion to Second Line Cervical Cancer
Brief Title: A Study of AGEN2034 in Advanced Tumors and Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-700-01
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Advanced Cancer; Cervical Cancer
Keywords: Antibodies; Immunologic effects; Physiological Effects of Drugs
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — balstilimab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Monotherapy (Experimental): Dose of 3 mg/kg intravenous (IV) every 2 weeks for up to 24 months.
  Interventions: Drug: AGEN2034

INTERVENTIONS:
Drug: AGEN2034 — Anti-programmed cell death protein-1 (PD-1) Monoclonal Antibody
  Other Names: Anti-PD-1

SUMMARY:
This is a 2-part trial: a Phase 1, open-label, dose-escalation study in participants with metastatic or locally advanced solid tumors, with a consecutive Phase 2 expansion to evaluate efficacy in participants with recurrent, unresectable, or metastatic (advanced) cervical cancer that has progressed after a platinum-based treatment regimen.

DETAILED DESCRIPTION:
Phase 1: Dose Escalation

Phase 1 will consist of a standard 3+3 dose escalation with the following escalating dose levels and schedules:

Part A1: 1, 3, and 10 milligrams/kilogram (mg/kg) administered every 2 weeks

Part A2: 6 and 10 mg/kg every 3 weeks

Each participant will stay on the dose level and schedule assigned at trial entry. Participants will receive AGEN2034 for a maximum of 2 years or until confirmed progression, unacceptable toxicity, or any criterion for stopping the study drug or withdrawal from the trial occurs.

A Safety Monitoring Committee (SMC) will assess safety; decide on dose-escalation and opening of backfill enrollment; define the recommended Phase 2 dose (RP2D); and determine opening of the Phase 2 cohorts.

In Part A1, the first participant of each cohort will be observed for 16 days (that is, ≥48 hours after second dose) for occurrence of dose-limiting toxicity (DLT) before the second participant is administered trial medication. Thereafter, within each cohort, consecutively enrolled participants may initiate treatment ≥48 hours after the prior enrolled participant-initiated treatment. Dose escalation will continue until the maximum tolerated dose (MTD) is reached or the maximum planned dose level (10.0 mg/kg) is shown to be safe. The MTD is defined as the dose below which ≥2 DLTs are observed.

Once Part A1 is completed, enrollment to Part A2 will begin. If <2 DLTs are observed in Part A1 at the maximum planned dose of 10 mg/kg every 2 weeks, open enrollment to Part A2 will begin with enrollment of 10 participants at 6 mg/kg every 3 weeks, followed by open enrollment of 10 participants at 10 mg/kg every 3 weeks. If ≥2 DLTs are observed in Part A1, at the maximum planned dose in Part A1, the standard 3+3 dose escalation will resume with Part A2 where consecutively enrolled participants in dose escalation may initiate treatment ≥48 hours after the prior enrolled participant-initiated treatment.

For cohorts in dose escalation, concurrent with the 3+3 dose escalation schema, additional participants will be backfilled to lower dose levels to ensure that each cohort enrolls a total of 10 participants. Participants enrolled to backfill cohorts may be enrolled simultaneously, without sequential dosing (that is, not required to wait 48 hours between 2 participants). These additional participants at each dose level will have the purpose of generating additional safety, pharmacokinetics, and receptor occupancy data, and will not undergo formal DLT observation.

Phase 2: Dose Expansion

To further characterize safety and efficacy, participants with recurrent, unresectable, or metastatic cervical cancer will be enrolled in Phase 2 and receive the RP2D of AGEN2034 (3 mg/kg every 2 weeks) for a maximum of 2 years or until confirmed progression, unacceptable toxicity, or any criterion for stopping the study drug or withdrawal from the trial occurs.

An SMC will assess safety, and an Independent Data Monitoring Committee will evaluate safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate by giving written informed consent. Participation in pharmacogenomics testing is optional.
2. Be ≥18 years of age.
3. Diagnosis and prior systemic treatment:

   1. Phase 1: Have a histologically or cytologically confirmed diagnosis of a metastatic or locally advanced solid tumor for which no standard therapy is available or standard therapy has failed.
   2. Phase 2: I. Have (1) a histologically or cytologically confirmed diagnosis of squamous-cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix, and (2) metastatic, locally advanced, and/or unresectable disease at the time of enrollment. Histologic confirmation of the original primary tumor is required via pathology report. Note: The following cervical tumors are not eligible: minimal deviation/adenoma malignum, gastric type adenocarcinoma, clear cell carcinoma, and mesonephric carcinoma. II. Has cervical cancer and has relapsed after a platinum-based treatment (first line) regimen for advanced (recurrent, unresectable, or metastatic) disease; Note: Participants who have received >1 prior systemic treatment regimen for their advanced or metastatic disease will be eligible in the following cases: Participant receiving chemotherapy concurrently with primary radiation (for example, weekly cisplatin) or participant receiving adjuvant chemotherapy following completion of radiation therapy (for example, paclitaxel and carboplatin for ≤4 cycles) and progressed within 6 months after treatment completion.
4. Measurable disease - based on investigator assessment

   1. Phase 1: Have objective evidence of disease; the presence of measurable disease is not required.
   2. Phase 2: Have measurable disease on imaging based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Note: Participants must have at least one "target lesion" to be used to assess response, as defined by RECIST 1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy. Note: Measurable disease by RECIST 1.1 must be confirmed by independent central radiologic review prior to first dose. Participants without centrally confirmed measurable disease at baseline will not be eligible for this trial.
5. Have a life expectancy of at least 3 months and an Eastern Cooperative Oncology Group performance status of 0 or 1.
6. Have adequate organ function as indicated by the following laboratory values:

   1. Adequate hematological function defined by absolute neutrophil count ≥1.5 x 10^9/liter (L), platelet count ≥100 x 10^9/L, and stable hemoglobin ≥8 grams/deciliter (without transfusions within 1 week before first dose).
   2. Adequate hepatic function based by a total bilirubin level ≤ the institutional upper limit of normal (IULN), aspartate aminotransferase level ≤2.5 x IULN, alanine aminotransferase level ≤2.5 x IULN, and alkaline phosphatase ≤2.5 x IULN.
   3. Adequate renal function defined as creatinine ≤1.5 x IULN or calculated creatinine clearance ≥50 milliliters/minute for participants with creatinine levels >1.5 x IULN (if no local guideline is available, creatinine clearance should be calculated using the Cockcroft-Gault Method).
   4. Adequate coagulation defined by international normalized ratio or prothrombin time ≤1.5 x IULN (unless the participant is receiving anticoagulant therapy); and activated partial thromboplastin time ≤1.5 x IULN (unless the participant is receiving anticoagulant therapy)
7. Other than the cancer for which the participant is enrolled, have no history of prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous-cell carcinoma of the skin, or has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
8. In Phase 2, participants must provide a sufficient and adequate formalin-fixed paraffin-embedded tumor tissue sample preferably from the most recent biopsy of a tumor lesion, collected either at the time of or after the diagnosis of advanced or metastatic disease has been made and from a site not previously irradiated. If no tumor tissue is available, a fresh biopsy will be required.

   Note: Tissue from needle or excisional biopsy or from resection is required.
9. Female participants must have a negative serum pregnancy test at screening (within 72 hours before first dose of study drug) if of childbearing potential or be of non-childbearing potential. Non-childbearing potential is defined as (by other than medical reasons):

   1. ≥45 years of age and has not menstruated for greater than 1 year,
   2. Amenorrheic for <2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation,
   3. Whose status is post hysterectomy, oophorectomy or tubal ligation.
10. If of childbearing potential, female participants must be willing to use 2 highly effective methods (defined in the informed consent form [ICF]) throughout the study, starting with the screening visit through 120 days after the last dose of study treatment.

    Note: Abstinence is acceptable if this is the established and preferred contraception for the participant.
11. Male participants with a female partner(s) of childbearing potential must agree to use 2 highly effective methods (defined in the ICF) throughout the trial starting with the screening visit through 120 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

    Note: Abstinence is acceptable if this is the established and preferred contraception for the participant.
12. Is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks before the first dose of treatment.
2. Has an inadequate washout period prior to first dose of study drug defined as:

   1. Received systemic cytotoxic chemotherapy or biological therapy within 3 weeks before first dose,
   2. Received radiation therapy within 3 weeks before first dose, or
   3. Had major surgery within 4 weeks before first dose.
3. Has received prior therapy with:

   1. Any antibody/drug targeting T-cell co-regulatory proteins (immune checkpoints) such as anti-PD-1, anti-programmed cell death ligand 1, or anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) antibodies
   2. For Phase 2: >1 systemic treatment regimen for the advanced (recurrent, unresectable, or metastatic) cervical cancer for which the participant is considered for the study Note: In Phase 1, prior treatment with a CTLA-4 antibody is permissible for participants with metastatic melanoma.
4. Has persisting toxicity related to prior therapy of National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE) Grade >1 severity.

   Note: Sensory neuropathy or alopecia of Grade ≤2 is acceptable.
5. Is expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
6. Has known severe hypersensitivity reactions to fully human monoclonal antibodies (NCI CTCAE Grade ≥3), any history of anaphylaxis, or uncontrolled asthma.
7. Is receiving systemic corticosteroid ≤7 days prior to the first dose of trial treatment or receiving any other form of systemic immunosuppressive medication (corticosteroid use on study for management of immune-related adverse events, and/or a premedication for IV contrast allergies/reactions is allowed). Participants who are receiving daily corticosteroid replacement therapy are an exception to this rule. Examples of permitted therapy are daily prednisone at doses of 5 to 7.5 mg or equivalent hydrocortisone dose, and steroid therapy administered by topical, intraocular, intranasal, and/or inhalation routes.
8. Has a central nervous system tumor, metastasis(es), and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period or identified prior to consent. Note: Participants with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions at screening (based on 2 sets of brain images, performed ≥4 weeks apart, and obtained after the brain metastases treatment). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be minimal and be expected as sequelae from treated lesions. For individuals who received steroids as part of brain metastases treatment, steroids must be discontinued ≥7 days prior to first dose of study drug.
9. Has active or history of autoimmune disease that has required systemic treatment within 2 years of the start of trial treatment (that is, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (that is, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Note: Participants with type 1 diabetes, vitiligo, psoriasis, hypo-, or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
10. Has had an allogeneic tissue/solid organ transplant.
11. Has or had interstitial lung disease or has had a history of pneumonitis that has required oral or IV corticosteroids.
12. Has an active infection requiring intravenous systemic therapy.
13. Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
14. Has known active Hepatitis B, Hepatitis C or tuberculosis. Active Hepatitis B is defined as a known positive Hepatitis B surface antigen result. Active Hepatitis C is defined by a known positive Hepatitis C antibody result and known quantitative Hepatitis C virus ribonucleic acid results greater than the lower limits of detection of the assay.
15. Has clinically significant (that is, active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months before enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥II), or serious uncontrolled cardiac arrhythmia requiring medication.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
19. Is legally incapacitated or has limited legal capacity.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (44):
- United States (12):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - University of Southern California - Keck School of Medicine, Los Angeles, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - Augusta Oncology, Augusta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Medical Center-Cherry Hill Campus, Seattle, Washington
- Australia (2):
  - Pindara Private Hospital, Benowa, Queensland
  - Calvary North Adelaide Hospital, North Adelaide, South Australia
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Brazil (7):
  - IMIP, Recife, Pernambuco
  - Instituto Nacional de Câncer, Rio de Janeiro, Rio de Janeiro
  - Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de São Paulo, São Paulo, São Paulo
  - Hospital Amaral Carvalho, São Paulo, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
- Chile (4):
  - Centro Oncológico del Norte, Antofagasta, AN
  - Centro De Investigación Del Cancer James Lind, Temuco, AR
  - Fundación Arturo López Pérez, Santiago, RM
  - Bradford Hill, Santiago, RM
- Estonia (2):
  - East-Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
- France (11):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - L'Institut Paoli - Calmettes, Marseille
  - CHU Hôpital de la Timone, Marseille
  - Centre Antoine-Lacassagne, Nice
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon - Hopital de la Croix Saint-Simon, Paris
  - Clinique Armoricaine de Radiologie, Plérin
  - Institute de Cancerologie de l'Ouest (ICO) - René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Poland (2):
  - Szpital Swietego Rafala w Krakowie, Krakow, Lesser Poland Voivodeship
  - Szpitale Pomorskie Sp. z o.o., Gdynia, Pomeranian Voivodeship
- Spain (3):
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Clínica Universidad de Navarra, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Balstilimab Dose 1: Participants received 1 milligram/kilogram (mg/kg) every 2 weeks (Q2W) balstilimab for up to 24 months.
- Phase 1: Balstilimab Dose 2: Participants received 3 mg/kg Q2W balstilimab for up to 24 months.
- Phase 1: Balstilimab Dose 3: Participants received 6 mg/kg every 3 weeks (Q3W) balstilimab for up to 24 months.
- Phase 1: Balstilimab Dose 4: Participants received 10 mg/kg Q2W balstilimab for up to 24 months.
- Phase 1: Balstilimab Dose 5: Participants received 10 mg/kg Q3W balstilimab for up to 24 months.
- Phase 2: Balstilimab Recommended Phase 2 Dose: Participants received 3 mg/kg Q2W balstilimab for a maximum of 24 months or until progression, unacceptable toxicity, stopping the study drug, or withdrawal from the study.
Period: Phase 1: Dose Escalation
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5 | Phase 2: Balstilimab Recommended Phase 2 Dose
Started | 10 | 10 | 10 | 10 | 10 | 0
Received at Least 1 Dose of Study Drug (Safety Analysis Set) | 10 | 10 | 10 | 10 | 10 | 0
Completed | 0 | 0 | 2 | 0 | 0 | 0
Not Completed | 10 | 10 | 8 | 10 | 10 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 4 | 8 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Death | 6 | 3 | 0 | 1 | 1 | 0
Not completed — Completed Follow Up | 2 | 2 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 0
Period: Phase 2: Dose Expansion
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5 | Phase 2: Balstilimab Recommended Phase 2 Dose
Started | 0 (Phase 1 participants did not continue into Phase 2.) | 0 (Phase 1 participants did not continue into Phase 2.) | 0 (Phase 1 participants did not continue into Phase 2.) | 0 (Phase 1 participants did not continue into Phase 2.) | 0 (Phase 1 participants did not continue into Phase 2.) | 161 (Phase 2 participants enrolled separately from Phase 1.)
Received at Least 1 Dose of Study Drug (Safety Analysis Set) | 0 | 0 | 0 | 0 | 0 | 161
Completed (Only deaths notified as leading to study discontinuation during Phase 2 are reported in the Participant Flow section. All deaths regardless of causality or whether they were reported as a reason for study discontinuation are reported in the All-Cause Mortality section.) | 0 | 0 | 0 | 0 | 0 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 133
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 107
Not completed — Participant Left to Participate in Another Trial | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Administrative Study Closure | 0 | 0 | 0 | 0 | 0 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of balstilimab.
Groups:
- Phase 1: Balstilimab Dose 1: Participants received 1 mg/kg Q2W balstilimab for up to 24 months.
- Phase 1: Balstilimab Dose 3: Participants received 6 mg/kg Q3W balstilimab for up to 24 months.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5 | Phase 2: Balstilimab Recommended Phase 2 Dose | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 161 | 211
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 7 | 9 | 6 | 7 | 6 | 119 | 154
  From 65-84 years | 3 | 1 | 4 | 3 | 4 | 42 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 9 | 9 | 8 | 161 | 203
  Male | 2 | 2 | 1 | 1 | 2 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 1 | 38 | 43
  Not Hispanic or Latino | 9 | 10 | 8 | 9 | 9 | 39 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 84 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 3 | 1 | 1 | 1 | 1 | 7
  Black or African American | 2 | 1 | 0 | 0 | 0 | 2 | 5
  White | 8 | 6 | 9 | 9 | 9 | 72 | 113
  Not Reported (France) | 0 | 0 | 0 | 0 | 0 | 81 | 81
  Romanian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Mixed | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Brown | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants Experiencing Dose-limiting Toxicities (DLTs) for Balstilimab
Description: A DLT was defined as any treatment-related toxicity that was National Cancer Institute Common Terminology Criteria for Adverse Event Grade ≥3, confirmed by the safety monitoring committee to be relevant for the study drug treatment, and that occurred during the first 3 weeks of balstilimab treatment in the dose escalation portion of the study (DLT evaluation period).
Time Frame: 21 days
Population: DLT Analysis Set: all participants who were enrolled for DLT evaluation (excluding participants enrolled to backfill cohorts) and either received all balstilimab administrations or stopped treatment due to a DLT during the DLT evaluation period. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which did not necessarily have a causal relationship with the treatment. TEAEs were AEs with onset dates during the on-treatment period, or the worsening of an event during the on-treatment period. A summary of all Serious Adverse Events and Other Adverse Events (nonserious), regardless of causality, is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 3 years
Population: Safety Analysis Set: all participants who received at least 1 dose of balstilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 10 | 10 | 10 | 10 | 10

3. Primary Outcome: Phase 2: Objective Response Rate (ORR) as Determined by an Independent Endpoint Review Committee (IERC)
Description: ORR was defined as percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR), as determined by an IERC per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). BOR was defined as the best response recorded from the start of the study treatment until the end of treatment. CR was defined as disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 3 years
Population: Intent-to-Treat Efficacy Analysis Set: all participants who received ≥1 dose of balstilimab with measurable disease at baseline (per IERC).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 160
percentage of participants | 15.6 [10.8 to 22.0]

4. Secondary Outcome: Phase 1: Receptor Occupancy of Circulating T Cells
Description: The percentage of PD-1 receptor occupancy on circulating T cells was measured as an indication of target engagement. An increase in percent occupancy indicates a potential increase in drug effectiveness.
Time Frame: 4 hours after the first dose (Cycle 1 Day 1) and immediately prior to the second dose (Cycle 2 Day 1) (2-3 weeks/cycle)
Population: Receptor Occupancy Analysis Set: all participants who completed ≥1 balstilimab infusion, with adequate measurements of PD-1 receptor occupancy on circulating T cells. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: percent occupancy
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5
Number analyzed (Participants) | 10 | 5 | 0 | 3 | 0
percent occupancy
  Cycle 1 Day 1 | 73.2 (11.95) | 69.4 (5.52) |  | 76.6 (2.95) |
  Cycle 2 Day 1: number analyzed (Participants) | 10 | 3 | 0 | 3 | 0
  Cycle 2 Day 1 | 67.7 (16.93) | 61.6 (1.70) |  | 72.1 (8.29) |

5. Secondary Outcome: Phase 1: Maximum Observed Concentration (Cmax) of Balstilimab
Description: Blood samples were collected for serum balstilimab concentration determinations. Results are reported as micrograms/milliliter (ug/mL).
Time Frame: Day 1 (Pre-dose up to 24 hours post dose) of Cycle 1 and Cycle 2 (2-3 weeks/cycle) (up to 3 weeks)
Population: Pharmacokinetic Analysis Set: all participants who completed ≥1 balstilimab infusion of study drug and who had sufficient evaluable drug concentration measurements prior to and after treatment. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10
ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 10 | 9 | 10 | 9 | 10
  Cycle 1 Day 1 | 18.1 (34.3) | 71.9 (19.5) | 153 (23.7) | 236 (26.6) | 282 (28.4)
  Cycle 2 Day 1: number analyzed (Participants) | 10 | 9 | 8 | 10 | 7
  Cycle 2 Day 1 | 20.3 (47.0) | 86.3 (30.0) | 161 (27.5) | 239 (28.2) | 315 (25.5)

6. Secondary Outcome: Phase 1: Area Under the Drug Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of Balstilimab
Description: Blood samples were collected for serum balstilimab concentration determinations. Results are reported as hours*micrograms/milliliter (h*µg/mL).
Time Frame: Day 1 (Pre-dose up to 24 hours post dose) of Cycle 1 and Cycle 2 (2-3 weeks/cycle) (up to 3 weeks)
Population: Pharmacokinetic Analysis Set: all participants who completed ≥1 balstilimab infusion and who had sufficient evaluable drug concentration measurements prior to and after treatment. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10
h*µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 10 | 9 | 10 | 9 | 10
  Cycle 1 Day 1 | 1265 (47.4) | 6470 (34.6) | 12632 (51.5) | 22294 (47.5) | 30751 (50.4)
  Cycle 2 Day 1: number analyzed (Participants) | 10 | 9 | 8 | 10 | 7
  Cycle 2 Day 1 | 1477 (73.7) | 7725 (40.2) | 17479 (49.4) | 21298 (47.1) | 42266 (41.0)

7. Secondary Outcome: Phase 1: Number of Participants With Serum Anti-drug Antibodies (ADAs) for Balstilimab
Description: Blood samples were collected for serum balstilimab ADA determination.
Time Frame: Up to 2.5 years
Population: Safety Analysis Set: all participants who received at least 1 dose of balstilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 3 | 0 | 0 | 0 | 0

8. Secondary Outcome: Phase 2: Number of Participants Experiencing TEAEs
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which did not necessarily have a causal relationship with the treatment. TEAEs were AEs with onset dates during the on-treatment period, or the worsening of an event during the on-treatment period. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 3 years
Population: Safety Analysis Set: all participants who received at least 1 dose of balstilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 161
Participants | 161

9. Secondary Outcome: Phase 2: Cmax of Balstilimab
Description: Blood samples were collected for serum balstilimab concentration determinations. Results are reported in μg/mL.
Time Frame: Day 1 (Pre-dose up to 24 hours post dose) of Cycle 1 and Cycle 2 (2 weeks/cycle) (up to 2 weeks)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 124
μg/mL
  Cycle 1 Day 1 | 55.4 (42.8)
  Cycle 2 Day 1: number analyzed (Participants) | 28
  Cycle 2 Day 1 | 56.6 (23.9)

10. Secondary Outcome: Phase 2: AUC0-last of Balstilimab
Description: Blood samples were collected for serum balstilimab concentration determinations. Results are reported in day*μg/mL.
Time Frame: Day 1 (Pre-dose up to 24 hours post dose) of Cycle 1 and Cycle 2 (2 weeks/cycle) (up to 2 weeks)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 124
day*μg/mL
  Cycle 1 Day 1 | 174 (46.3)
  Cycle 2 Day 1: number analyzed (Participants) | 28
  Cycle 2 Day 1 | 184 (59.7)

11. Secondary Outcome: Phase 2: Number of Participants With Serum ADAs for Balstilimab
Description: Blood samples were collected for serum balstilimab ADA determination.
Time Frame: Up to 2.5 years
Population: Safety Analysis Set: all participants who received at least 1 dose of balstilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 161
Participants | 7

12. Secondary Outcome: Phase 2: ORR as Determined by the Investigator
Description: ORR was defined as percentage of participants with a BOR of CR or PR, as determined by the investigator per RECIST 1.1. BOR was defined as the best response recorded from the start of the study treatment until the end of treatment. CR was defined as disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 3 years
Population: Intent-to-Treat Efficacy Analysis Set: all participants who received ≥1 dose of balstilimab with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 160
percentage of participants | 14.4 [9.8 to 20.6]

13. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was defined as time from first observation of response to first observation of documented progressive disease (PD) (or death within 12 weeks after last tumor assessment), per RECIST 1.1 and as determined by an IERC and the investigator. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). Participants without an event at analysis cutoff date were censored on date of last tumor assessment.
Time Frame: Up to 3 years
Population: Intent-to-Treat Efficacy Analysis Set: all participants who received ≥1 dose of balstilimab with measurable disease at baseline (per IERC). Here, 'Overall Number of Participants Analyzed' and 'Number Analyzed' signify those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 25
months
  IERC | NA [7.3 to NA] — The upper bound of the 95% confidence interval of the median could not be estimated as the median was not reached at the data cut-off.
  Investigator: number analyzed (Participants) | 23
  Investigator | NA [8.9 to NA] — The upper bound of the 95% confidence interval of the median could not be estimated as the median was not reached at the data cut-off.

14. Secondary Outcome: Phase 2: Disease Control Rate (DCR) as Determined by an IERC
Description: DCR was defined as the percentage of participants with CR, PR, or stable disease (SD) for at least 12 weeks. CR was defined as disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study).
Time Frame: Up to 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 160
percentage of participants | 50.6 [43.0 to 58.3]

15. Secondary Outcome: Phase 2: Tumor Control Rate (TCR) as Determined by an IERC
Description: TCR was defined as percentage of participants who had a BOR of either SD or a confirmed objective response (CR or PR). CR was defined as disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study).
Time Frame: Up to 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 160
percentage of participants | 52.5 [44.8 to 60.1]

16. Secondary Outcome: Phase 2: Time to Response (TTR) as Determined by an IERC
Description: TTR was defined as the time from the first dose date to first observation of confirmed response.
Time Frame: Up to 3 years
Population: Intent-to-Treat Efficacy Analysis Set: all participants who received ≥1 dose of balstilimab with measurable disease at baseline (per IERC). Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 25
days | 82.0 [60.5 to 108.4]

17. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as time from first treatment administration to first observation of documented PD (or death within 12 weeks after last tumor assessment), per RECIST 1.1, as determined by an IERC and investigator. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). Participants without an event at analysis cutoff date were censored on date of last tumor assessment.
Time Frame: Up to 3 years
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 137
months
  IERC: number analyzed (Participants) | 132
  IERC | 2.8 [2.4 to 3.9]
  Investigator | 3.6 [2.7 to 4.2]

18. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as time from start of treatment to death. For participants who were still alive at the time of data cutoff for trial analysis or who were lost to follow-up, survival was censored at the last recorded date that the participant was known to have been alive as of the cutoff date for analysis.
Time Frame: Up to 3 years
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Balstilimab Recommended Phase 2 Dose
Number analyzed (Participants) | 108
months | 11.2 [9.5 to 14.5]

ADVERSE EVENTS:
Time Frame: From Day 1 to the end of study (3 years)
Description: All reported safety data based upon the Safety Analysis Set: all participants who received at least 1 dose of balstilimab.
  All deaths regardless of causality or whether they were reported as a reason for study discontinuation are reported in the All-Cause Mortality section. Only deaths notified as leading to study discontinuation during Phase 2 are reported in the Participant Flow section.
Arm/Group | Phase 1: Balstilimab Dose 1 | Phase 1: Balstilimab Dose 2 | Phase 1: Balstilimab Dose 3 | Phase 1: Balstilimab Dose 4 | Phase 1: Balstilimab Dose 5 | Phase 2: Balstilimab Recommended Phase 2 Dose
All-Cause Mortality (participants affected / at risk) | 6/10 | 3/10 | 0/10 | 1/10 | 1/10 | 108/161
Serious Adverse Events (participants affected / at risk) | 5/10 | 3/10 | 5/10 | 3/10 | 2/10 | 90/161
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 10/10 | 10/10 | 158/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Phase 1: Balstilimab Dose 1 (N=10) | Phase 1: Balstilimab Dose 2 (N=10) | Phase 1: Balstilimab Dose 3 (N=10) | Phase 1: Balstilimab Dose 4 (N=10) | Phase 1: Balstilimab Dose 5 (N=10) | Phase 2: Balstilimab Recommended Phase 2 Dose (N=161)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 5
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 4
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/8 | 0/8 | 0/9 | 0/9 | 0/8 | 3 — This is a sex-specific adverse event. Only female participants were at risk.
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0/8 | 0/8 | 0/9 | 0/9 | 0/8 | 1 — This is a sex-specific adverse event. Only female participants were at risk.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Aortic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Upper GI haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 7
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 6
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Postrenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urogenital fistula (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Arboviral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Phase 1: Balstilimab Dose 1 (N=10) | Phase 1: Balstilimab Dose 2 (N=10) | Phase 1: Balstilimab Dose 3 (N=10) | Phase 1: Balstilimab Dose 4 (N=10) | Phase 1: Balstilimab Dose 5 (N=10) | Phase 2: Balstilimab Recommended Phase 2 Dose (N=161)
Nausea (Gastrointestinal disorders) | 6 | 3 | 4 | 5 | 3 | 47
Constipation (Gastrointestinal disorders) | 4 | 2 | 2 | 1 | 1 | 45
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 2 | 3 | 2 | 41
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2 | 5 | 1 | 38
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 3 | 2 | 35
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 11
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 1 | 56
Fatigue (General disorders) | 7 | 4 | 3 | 7 | 3 | 37
Pyrexia (General disorders) | 0 | 0 | 3 | 3 | 1 | 35
Oedema peripheral (General disorders) | 0 | 1 | 1 | 1 | 1 | 21
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 3 | 3 | 3 | 80
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 3 | 2 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 1 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 1 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 9
Urinary tract infection (Infections and infestations) | 2 | 3 | 0 | 0 | 3 | 35
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 3 | 5 | 2 | 34
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 10
Blood creatinine increased (Investigations) | 1 | 2 | 1 | 0 | 0 | 17
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 17
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 2 | 2 | 0 | 17
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 2 | 16
Weight decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 16
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 13
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 3 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 0 | 2 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 30
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 9
Headache (Nervous system disorders) | 1 | 1 | 1 | 3 | 1 | 26
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 10
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 9
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 9
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 25
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/8 | 0/8 | 0/9 | 0/9 | 0/8 | 16 — This is a sex-specific adverse event. Only female participants were at risk.
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 16
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 0 | 0 | 15
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 11
Immune-mediated hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 9
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 8
Ascites (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 6
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 4
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lip erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 7
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 1 | 0 | 4
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 3
Oedema (General disorders) | 1 | 0 | 0 | 0 | 1 | 2
Malaise (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 3 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 5
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 4
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 4
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 5
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 2 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 2 | 2 | 1 | 8
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 7
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 5
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 6
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 2
Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0/2 | 1/2 | 0/1 | 1/1 | 0/2 | 0/0 — This is a sex-specific adverse event. Only male participants were at risk.
Vaginal odour (Reproductive system and breast disorders) | 0/8 | 0/8 | 0/9 | 0/9 | 1/8 | 0 — This is a sex-specific adverse event. Only female participants were at risk.
Depression (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0 | 6
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 3
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 4
Flushing (Vascular disorders) | 0 | 0 | 2 | 1 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 2
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Stoma site irritation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT03104699/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT03104699/SAP_001.pdf